CLINICAL TRIAL: NCT04975386
Title: Echocardiographic Investigation of the Cardiac Effects of Different Regional Anesthesia Methods Used in Intertrochanteric Femoral Fracture Operations
Brief Title: Echocardiography Examination Of The Cardiac Effects Of Different Regional Anesthesia Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator ,Assoc. PhD. M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25 2020/10-03
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Femur Fracture; Spinal Anesthesia; Lumbar Plexus Block
MeSH Terms: conditions — Femoral Fractures | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal anesthesia (Active Comparator)
  Interventions: Device: Transthoracic echocardiogram
- lumbar plexus+sacral plexus block (Active Comparator)
  Interventions: Device: Transthoracic echocardiogram

INTERVENTIONS:
Device: Transthoracic echocardiogram — Transthoracic echocardiogram will be performed before the operation and at certain time intervals during the operation.

SUMMARY:
Nerve blocks applied with neuraxial anesthesia and ultrasonography are used for many operations today. Neuraxial blocks cause varying degrees of decrease in the blood pressure level of the patients. Peripheral blocks may be preferred to avoid the cardiac effects of the neuraxial anesthesia method.

DETAILED DESCRIPTION:
The hypothesis of this study was that spinal anesthesia applied in intertrochanteric femoral fracture operations caused hypotension by lowering the cardiac ejection fraction.

In our study, The investigators aimed to find out the effect of different regional anesthesia methods on the cardiac function of the patients by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* 60-100 years old
* American Society of Anesthesiologist Score I-IV

Exclusion Criteria:

* Local anesthetic allergy
* Bleeding disorder
* Mental disorder
* Allergy to drugs used
* Body mass index above 30

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-07-29 (Estimated); Primary Completion 2022-07-29 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Ejection fraction | peroperative
  Ejection fraction (EF) measurement will be made with Simpson's method and fractional shortening method.

SECONDARY OUTCOMES:
intraoperative blood pressure monitoring | peroperative
  systolic, diastolic and median blood pressure values
cardiac diastolic dysfunction | peroperative
  The echocardiogram will measure the flow velocity between the left atrium and ventricle in cm/s in pulsed wave mode and the E/A ratio will be calculated.
Entropy | peroperative
  Depth of anesthesia will be measured by placing Entropy sensors on the forehead as needed.
sedative drug | intraoperative
  The drugs used for sedation and their amounts will be recorded.
ramsey sedation scale | intraoperative
  1. point Awake, restless and/or crying.
  2. points Alert, calm, watching his surroundings.
  3. points Sleepy but responds to verbal stimuli
  4. points Sleepy but immediately responds to glabellar tactile stimuli.
  5. points Sleepy but responds slowly to glabellar tactile stimuli.
  6. points Does not respond to Alerts.

CONTACTS AND LOCATIONS:
Overall Officials: Durdu M.D Kahraman Yıldız, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No